CLINICAL TRIAL: NCT06054971
Title: Use of Telemedicine and At-Home Video for Remote Administration of the North Star Ambulatory Assessment (NSAA): a Feasibility Study
Brief Title: NSAA NON-Interventional Study Protocol
Status: Completed | Type: Observational
Sponsor: Red Nucleus Enterprise Solutions, LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Christopher Jones, PhD, Principal Investigator, Red Nucleus Enterprise Solutions, LLC
Other Study IDs: NSAA-RWE-001
Record Dates: First submitted 2023-09-12; First posted 2023-09-26 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-11

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: Group A will have Live telemedicine assessments completed prior to caregiver Asynchronous Video
  Interventions: Other: Remote Administration of NSAA
- Group B: Group B will have Caregiver Asynchronous Video first, followed by live telemedicine
  Interventions: Other: Remote Administration of NSAA

INTERVENTIONS:
Other: Remote Administration of NSAA — Remote Administration of NSAA

SUMMARY:
The purpose of this non-interventional study is to evaluate the feasibility of remotely administering the North Star Ambulatory Assessment (NSAA) to participants with Duchenne muscular dystrophy (DMD). The iTakeControl (iTC) software platform will be utilized to remotely administer and score the NSAAs.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a signed and dated informed consent document indicating that the participant's legally authorized representative (LAR) has been informed of all pertinent aspects of the study, along with evidence of age-appropriate child assent.
2. Confirmed diagnosis of DMD
3. Participant with DMD aged 4 to12 (inclusive) at t Enrollment date
4. Participant with DMD is ambulatory without assistive devices, braces, or aids throughout the study
5. Caregiver has access to and/or willingness to learn use of a smart phone and the iTC study mobile application
6. Participant and caregiver are based in the US throughout study
7. Participant and caregiver are fluent in the English language (verbally and in writing)

Exclusion Criteria:

1. Non-ambulatory DMD participant at any study timepoint
2. Caregiver/participant unwilling or unable to administer/perform the NSAA
3. Anticipated deterioration of participant's ambulatory status during the study

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Individuals with confirmed diagnosis of DMD
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Comparison of performance and ratings of the NSAA using three methods: 1) Live Telemedicine scores 2) Subsequent Recorded Telemedicine scores 3) Caregiver Asynchronous Video scores | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Red Nucleus Solutions, Malvern, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No